CLINICAL TRIAL: NCT03353415
Title: Determining the Efficacy of Continuous Glucose Monitoring to Reduce Hypoglycemia and Improve Safety in Patients With Hypoglycemia After Gastric Surgery
Brief Title: Continuous Glucose Monitoring to Reduce Hypoglycemia and Improve Safety After Gastric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joslin Diabetes Center (Other)
Collaborators: DexCom, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2017-27
Record Dates: First submitted 2017-11-21; First posted 2017-11-27 (Actual); Results first posted 2023-08-14 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Hypoglycemia, Reactive; Hypoglycemia
Keywords: Post-bariatric Hypoglycemia;
MeSH Terms: conditions — Hypoglycemia

STUDY DESIGN:
Intervention Model Description: The proposed study is designed to assess the efficacy of unmasked personal CGM to reduce the frequency of hypoglycemia after gastric surgery. Specifically, we will analyze glycemic patterns during a phase of baseline masked CGM wear (2 weeks for the Dexcom G4 or 10 days for the Dexcom G6), in comparison to a sequential, second phase of unmasked CGM wear (2 weeks for the Dexcom G4 or 10 days for the Dexcom G6). Please note that we have chosen to have a consistent masked monitoring first, as providing unmasked data to participants first could alter their dietary or other patterns and reduce ability of the study to independently assess efficacy of the CGM intervention.
Masking Description: The proposed study is designed to assess the efficacy of unmasked personal CGM to reduce the frequency of hypoglycemia after gastric surgery. Participants themselves will not be masked to study design. The only masking will be of the device sensor glucose data during the first 2 weeks (Dexcom G4) or 10 days (Dexcom G6) of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Masked CGM Wear (Phase 1) (Other): Each participant will wear the Dexcom CGM for two sequential phases. During the first phase, participants will not be able to read the sensor glucose levels (masked).
  Interventions: Device: Dexcom CGM masked
- Unmasked CGM Wear (Phase 2) (Experimental): In the second phase, participants will be able to read the sensor glucose levels (unmasked). Frequency of hypoglycemia will be compared between the two phases of the study.
  Interventions: Device: Dexcom CGM unmasked

INTERVENTIONS:
Device: Dexcom CGM masked — The CGM will monitor sensor glucose levels in all participants. (Initially the Dexcom G4 was worn by participants (n=13); however, when the G4 became unavailable, the G6 was worn by the subsequent participants (n=10)).
  The duration of the Dexcom G4 sensor was 7 days (2 sensors placed during each phase of participation) versus the Dexcom G6 whose sensor duration is 10 days (1 sensor placed during each phase of participation).
  Arms: Masked CGM Wear (Phase 1)
Device: Dexcom CGM unmasked — During the second phase (2 weeks for the Dexcom G4 and 10 days for the Dexcom G6), participants are able to see the sensor glucose levels displayed from the CGM. Participants will be instructed to use this information to treat low glucose levels before symptoms or severely low glucose levels develop.
  The duration of the Dexcom G4 sensor was 7 days (2 sensors placed during each phase of participation) versus the Dexcom G6 whose sensor duration is 10 days (1 sensor placed during each phase of participation).
  Arms: Unmasked CGM Wear (Phase 2)

SUMMARY:
The purpose of this study is to see if the use of a continuous glucose monitor (CGM) by people who experience low blood sugars (hypoglycemia) after gastric surgery can help reduce the number and severity of low blood sugar episodes.

DETAILED DESCRIPTION:
The CGM devices used in this study are approved by the Food and Drug Administration (FDA) for monitoring the glucose levels of people with diabetes. The investigators of this study are looking to see if these CGM devices are able to benefit people who have had gastric surgery and experience low blood sugar episodes, which can be asymptomatic and lead to complications, impairing safety. This study involves wearing a CGM sensor/transmitter during first a masked phase (unable to see CGM sensor glucose levels), followed by an unmasked phase (able to see and respond to sensor glucose levels and alarms). Participants are asked to regularly record fingerstick (capillary) blood sugar values and any symptoms experienced, as well as a record of treatments for symptoms and glucose levels.

Participants attend three to five study visits: 5 visits for participants who wore the Dexcom G4, and 3 visits for participants who wore the Dexcom G6. The Dexcom G4 became unavailable during the course of the study when the G6 was introduced. (The Dexcom G4 had a 7 day wear period versus a 10 day wear period for the G6. As the G6 has a longer wear period, the frequency of the study visits was able to be decreased).

This study also involves the use of a fitness tracker, which will be worn for the duration of the study and returned at the end of the study.

Participants wearing the Dexcom G4 device were able to keep the Dexcom G4 CGM receiver and transmitter (this was not possible with the Dexcom G6 system).

ELIGIBILITY:
Inclusion Criteria:

1. Males or females diagnosed with ongoing post-bariatric or post-gastric surgery hypoglycemia with prior episodes of neuroglycopenia
2. Age 18-65 years of age, inclusive, at screening
3. Willingness to provide informed consent and follow all study procedures, including attending all scheduled visits.

Exclusion Criteria:

1. Documented hypoglycemia occurring in the fasting state (> 12 hours fast);
2. Chronic kidney disease stage 4 or 5 (including end-stage renal disease);
3. Hepatic disease, including serum alanine transaminase (ALT) or aspartate aminotransferase (AST) greater than or equal to 3 times the upper limit of normal; hepatic synthetic insufficiency as defined as serum albumin < 3.0 g/dL; or serum bilirubin >2.0;
4. Congestive heart failure, New York Heart Association (NYHA) class II, Ill or IV;
5. History of myocardial infarction, unstable angina or revascularization within the past 6 months or 2 or more risk factors for coronary artery disease including diabetes, uncontrolled hypertension, uncontrolled hyperlipidemia, and active tobacco use.
6. History of syncope (unrelated to hypoglycemia) or diagnosed cardiac arrhythmia
7. Concurrent administration of beta-blocker therapy;
8. History of a cerebrovascular accident;
9. Seizure disorder (other than with suspect or documented hypoglycemia);
10. Active treatment with any diabetes medications except for acarbose;
11. Active treatment with octreotide or diazoxide;
12. Active malignancy, except basal cell or squamous cell skin cancers;
13. Personal or family history of pheochromocytoma or disorder with increased risk of pheochromocytoma (multiple endocrine neoplasia (MEN) 2, neurofibromatosis, or Von Hippel-Lindau disease);
14. Known insulinoma;
15. Major surgical operation within 30 days prior to screening;
16. Hematocrit< 33%;
17. Bleeding disorder, treatment with warfarin, or platelet count <50,000;
18. Blood donation (1 pint of whole blood) within the past 2 months;
19. Active alcohol abuse or substance abuse;
20. Current administration of oral or parenteral corticosteroids;
21. Pregnancy and/ or lactation: For women of childbearing potential: there is a requirement for a negative urine pregnancy test and for agreement to use contraception during the study and for at least 1 month after participating in the study. Acceptable contraception includes birth control pill/patch I vaginal ring, Depo-Provera, Norplant, an intrauterine device (IUD), the double barrier method (the woman uses a diaphragm and spermicide and the man uses a condom), or abstinence.
22. Use of an investigational drug within 30 days prior to screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-02-07 (Actual); Primary Completion 2021-11-11 (Actual); Study Completion 2023-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Elizabeth Patti, MD, Principal Investigator — Joslin Diabetes Center
Locations (1):
- Joslin Diabetes Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Patti ME, Goldfine AB. The rollercoaster of post-bariatric hypoglycaemia. Lancet Diabetes Endocrinol. 2016 Feb;4(2):94-6. doi: 10.1016/S2213-8587(15)00460-X. Epub 2015 Dec 15. No abstract available. PMID 26701701
- [Result] Cummings C, Jiang A, Sheehan A, Ferraz-Bannitz R, Puleio A, Simonson DC, Dreyfuss JM, Patti ME. Continuous glucose monitoring in patients with post-bariatric hypoglycaemia reduces hypoglycaemia and glycaemic variability. Diabetes Obes Metab. 2023 Aug;25(8):2191-2202. doi: 10.1111/dom.15096. Epub 2023 May 3. PMID 37046360

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with post-gastric surgery hypoglycemia were recruited from the Hypoglycemia Clinic at Joslin Diabetes Center, directed by Dr. Patti. The study was explained to potential participants initially in the clinical setting or during a subsequent telephone screening session.
  Recruitment took place between February of 2019 through December of 2021. The dexcom G4 was available for the first 13 participants. The remaining 10 participants wore the dexcom G6.
Pre-assignment Details: After enrollment, 1 participant was withdrawn and did not complete baseline evaluation (visit 1) due to hospitalization.
  Following baseline evaluation (visit 1), 2 participants were lost to followup and did not complete the masked CGM wear period.
  One additional participant was excluded due to missing data and therefore could not be included in the analyses.
Groups:
- CGM Use: Each participant wore the Dexcom continuous glucose monitor (CGM) available at their time of participation. The Dexcom G4 became unavailable during the course of the study and later participants wore the Dexcom G6. During the first two weeks (Dexcom G4) or first 10 days (Dexcom G6), participants were not able to read the sensor glucose levels. In the second two weeks (Dexcom G4) or second 10 days (Dexcom G6), participants were able to read the sensor glucose levels. Frequency of hypoglycemia was compared between the two phases of the study (masked versus unmasked CGM).
  Dexcom CGM: The CGM monitored sensor glucose levels in all participants. During the first two weeks (Dexcom G4) or first 10 days (Dexcom G6) of the study, participants were masked to the sensor glucose levels and needed to use other methods, such as a blood sample from a finger stick, to check their blood sugar. During the second two weeks (Dexcom G4) or second10 days (Dexcom G6), participants were able to see the sensor glucose levels displayed from the CGM. Participants were instructed to use this information to treat low glucose levels before symptoms or severely low glucose levels developed.
Period: Masked CGM Wear
Arm/Group | CGM Use
Started (26 individuals were enrolled, however one individual was withdrawn prior to participation due to hospitalization. No study visits were attended or study related activities initiated for this person. 25 participants completed the visit 1 baseline evaluation.) | 25
Completed | 23
Not Completed | 2
Not completed — Lost to Follow-up | 2
Period: Unmasked CGM Wear
Arm/Group | CGM Use
Started | 23
Completed | 22
Not Completed | 1
Not completed — Excluded due to missing data. | 1

BASELINE CHARACTERISTICS:
Population: 25 participants completed baseline evaluation after enrollment and these are reflected in this analysis. After baseline evaluation 2 participants were lost to follow-up before CGM download, and 1 participant's CGM data was corrupted; therefore all analysis after baseline assessment are for a total of 22 participants.
Arm/Group | CGM Use
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.1 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 22
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25
Hemoglobin A1c [Mean (Standard Deviation); unit: percent] | 5.3 (0.4)
Pre-operative Body Mass Index (BMI) [Mean (Standard Deviation); unit: mg/k^2] | 47.6 (6.4)
Current BMI [Mean (Standard Deviation); unit: mg/k^2] | 30.6 (6.1)
Years post-bariatric surgery [Mean (Standard Deviation); unit: years] | 9.6 (8.1)
Years between bariatric surgery and hypoglycemia onset [Mean (Standard Deviation); unit: years] | 4.7 (6.3)
Percentage of participants with a history of level III hypoglycemia (requiring assistance) [Number; unit: percentage of participants] | 84
Percentage of participants with a history of neuroglycopenia [Number; unit: percentage of participants] | 100
Visit 1 Edinburgh Hypoglycemia Symptom Scale (EHSS) Score [Mean (Standard Deviation); unit: units on a scale (EHSS score)] — EHSS score range 18 to 126, with a higher number indicating a greater symptom severity score.
  units on a scale (EHSS score) | 49.3 (20.5)
Visit 1 Dumping Symptom Rating Scale (DSRS) Score [Mean (Standard Deviation); unit: units on a scale (DSRS score)] — DSRS scores range 9 to 56, with a higher score indicating a greater symptom severity score.
  units on a scale (DSRS score) | 23.1 (7.4)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Time Sensor Glucose <70 mg/dL in the Masked Versus the Unmasked Phase.
Description: The primary outcome will be time spent in hypoglycemic glucose range as measured by percent time sensor glucose is <70 mg/dl, comparing the masked versus the unmasked phases.
Time Frame: 28 days for those participants wearing Dexcom G4, and 20 days for participants wearing Dexcom G6.
Measure: Median (Standard Deviation); unit: Percentage of time
Groups:
- Masked CGM Wear (Phase 1): During the first phase, participants will not be able to read the sensor glucose levels (masked).
  Dexcom CGM masked: The CGM will monitor sensor glucose levels in all participants. (Initially the Dexcom G4 was worn by participants (n=13); however, when the G4 became unavailable, the G6 was worn by the subsequent participants (n=10)).
  The duration of the Dexcom G4 sensor was 7 days (2 sensors placed during each phase of participation) versus the Dexcom G6 whose sensor duration is 10 days (1 sensor placed during each phase of participation).
- Unmasked CGM Wear (Phase 2): During the second phase, participants will be able to read the sensor glucose levels (unmasked). Participants will be instructed to use this information to treat low glucose levels before symptoms or severely low glucose levels develop.
  The duration of the Dexcom G4 sensor was 7 days (2 sensors placed during each phase of participation) versus the Dexcom G6 whose sensor duration is 10 days (1 sensor placed during each phase of participation).
Arm/Group | Masked CGM Wear (Phase 1) | Unmasked CGM Wear (Phase 2)
Number analyzed (Participants) | 22 | 22
Percentage of time | 4.7 (4.8) | 2.9 (2.5)
Statistical Analysis 1: Comparison: Masked CGM Wear (Phase 1) vs Unmasked CGM Wear (Phase 2); Test type: Other; p = 0.04, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Percentage of Time Sensor Glucose <60mg/dL in the Masked Versus the Unmasked Phase
Description: The primary outcome will be time spent in hypoglycemic glucose range as measured by percent time sensor glucose is <60 mg/dl, comparing the masked versus the unmasked phases.
Time Frame: 28 days for those participants wearing Dexcom G4, and 20 days for participants wearing Dexcom G6.
Measure: Median (Standard Deviation); unit: Percentage of time
Arm/Group | Masked CGM Wear (Phase 1) | Unmasked CGM Wear (Phase 2)
Number analyzed (Participants) | 22 | 22
Percentage of time | 1.4 (1.7) | 0.7 (0.8)
Statistical Analysis 1: Comparison: Masked CGM Wear (Phase 1) vs Unmasked CGM Wear (Phase 2); Test type: Other; p = 0.03, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Percentage of Time Sensor Glucose <54 mg/dL in the Masked Versus the Unmasked Phase
Description: as for outcome 2
Time Frame: 28 days for those participants wearing Dexcom G4, and 20 days for participants wearing Dexcom G6.
Measure: Median (Standard Deviation); unit: Percentage of time
Arm/Group | Masked CGM Wear (Phase 1) | Unmasked CGM Wear (Phase 2)
Number analyzed (Participants) | 22 | 22
Percentage of time | 0.6 (0.8) | 0.2 (0.3)
Statistical Analysis 1: Comparison: Masked CGM Wear (Phase 1) vs Unmasked CGM Wear (Phase 2); Test type: Other; p = 0.14, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Median Sensor Glucose Level During Masked Versus Unmasked Phases of Wear
Time Frame: 28 days for those participants wearing Dexcom G4, and 20 days for participants wearing Dexcom G6.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Masked CGM Wear (Phase 1) | Unmasked CGM Wear (Phase 2)
Number analyzed (Participants) | 22 | 22
mg/dL | 97.5 [87.0 to 113.5] | 97.0 [87.0 to 113.0]
Statistical Analysis 1: Comparison: Masked CGM Wear (Phase 1) vs Unmasked CGM Wear (Phase 2); Test type: Other; p = 0.45, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Mean Sensor Glucose Level During Masked Versus Unmasked Phases of Wear
Time Frame: 28 days for those participants wearing Dexcom G4, and 20 days for participants wearing Dexcom G6.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Masked CGM Wear (Phase 1) | Unmasked CGM Wear (Phase 2)
Number analyzed (Participants) | 22 | 22
mg/dL | 103.8 (12.3) | 104.1 (7.4)
Statistical Analysis 1: Comparison: Masked CGM Wear (Phase 1) vs Unmasked CGM Wear (Phase 2); Test type: Other; p = 0.35, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Peak Sensor Glucose Level During Masked Versus Unmasked Period of CGM Wear
Description: expressed as median and median standard deviation
Time Frame: 28 days for those participants wearing Dexcom G4, and 20 days for participants wearing Dexcom G6.
Measure: Median (Standard Deviation); unit: mg/dL
Arm/Group | Masked CGM Wear (Phase 1) | Unmasked CGM Wear (Phase 2)
Number analyzed (Participants) | 22 | 22
mg/dL | 263.0 (51.9) | 256.0 (42.3)
Statistical Analysis 1: Comparison: Masked CGM Wear (Phase 1) vs Unmasked CGM Wear (Phase 2); Test type: Other; p = 0.53, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Sensor Glucose Level Range (Highest Sensor Glucose Minus Lowest Sensor Glucose mg/dL) During Masked Versus Unmasked Period of CGM Wear
Description: The sensor glucose level range is derived from the difference between the highest sensor glucose levels minus the lowest sensor glucose level (mg/dL).
Time Frame: 28 days for those participants wearing Dexcom G4, and 20 days for participants wearing Dexcom G6.
Measure: Median (Standard Deviation); unit: mg/dL
Arm/Group | Masked CGM Wear (Phase 1) | Unmasked CGM Wear (Phase 2)
Number analyzed (Participants) | 22 | 22
mg/dL | 221.5 (52.6) | 209.5 (50.4)
Statistical Analysis 1: Comparison: Masked CGM Wear (Phase 1) vs Unmasked CGM Wear (Phase 2); Test type: Other; p = 0.47, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Nadir Sensor Glucose Level During Masked Versus Unmasked Period of CGM Wear
Time Frame: 28 days for those participants wearing Dexcom G4, and 20 days for participants wearing Dexcom G6.
Measure: Median (Standard Deviation); unit: mg/dL
Arm/Group | Masked CGM Wear (Phase 1) | Unmasked CGM Wear (Phase 2)
Number analyzed (Participants) | 22 | 22
mg/dL | 40.0 (0.0) | 42.0 (3.0)
Statistical Analysis 1: Comparison: Masked CGM Wear (Phase 1) vs Unmasked CGM Wear (Phase 2); Test type: Other; p = 0.65, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Percent of Time Sensor Glucose 70-180 mg/dL During Period of CGM Wear, Masked Versus Unmasked Phase
Time Frame: 28 days for those participants wearing Dexcom G4, and 20 days for participants wearing Dexcom G6.
Measure: Median (Standard Deviation); unit: Percentage of time
Arm/Group | Masked CGM Wear (Phase 1) | Unmasked CGM Wear (Phase 2)
Number analyzed (Participants) | 22 | 22
Percentage of time | 90.8 (5.2) | 94.8 (3.9)
Statistical Analysis 1: Comparison: Masked CGM Wear (Phase 1) vs Unmasked CGM Wear (Phase 2); Test type: Other; p = 0.004, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Percentage of Time Sensor Glucose Level >180 mg/dL During Period of CGM Wear, Masked Versus Unmasked Phase
Time Frame: 28 days for those participants wearing Dexcom G4, and 20 days for participants wearing Dexcom G6.
Measure: Median (Standard Deviation); unit: Percentage of time
Arm/Group | Masked CGM Wear (Phase 1) | Unmasked CGM Wear (Phase 2)
Number analyzed (Participants) | 22 | 22
Percentage of time | 3.1 (2.8) | 1.7 (1.6)
Statistical Analysis 1: Comparison: Masked CGM Wear (Phase 1) vs Unmasked CGM Wear (Phase 2); Test type: Other; p = 0.05, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Percentage of Time Sensor Glucose Level >250 mg/dL During Periods of CGM Wear, Masked Versus Unmasked Phase
Time Frame: 28 days for those participants wearing Dexcom G4, and 20 days for participants wearing Dexcom G6.
Measure: Median (Standard Deviation); unit: Percentage of time
Arm/Group | Masked CGM Wear (Phase 1) | Unmasked CGM Wear (Phase 2)
Number analyzed (Participants) | 22 | 22
Percentage of time | 0.1 (0.2) | 0.1 (0.1)
Statistical Analysis 1: Comparison: Masked CGM Wear (Phase 1) vs Unmasked CGM Wear (Phase 2); Test type: Other; p = 0.22, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Glycemic Variability as Measured by the Standard Deviation of Sensor Glucose Level Data During Periods of CGM Wear, Masked Versus Unmasked Phase
Time Frame: 28 days for those participants wearing Dexcom G4, and 20 days for participants wearing Dexcom G6.
Measure: Median (Standard Deviation); unit: mg/dL
Arm/Group | Masked CGM Wear (Phase 1) | Unmasked CGM Wear (Phase 2)
Number analyzed (Participants) | 22 | 22
mg/dL | 29.8 (7.1) | 26.6 (5.2)
Statistical Analysis 1: Comparison: Masked CGM Wear (Phase 1) vs Unmasked CGM Wear (Phase 2); Test type: Other; p = 0.09, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: Mean Coefficient of Variation of Sensor Glucose Data During Period of CGM Wear, Masked Versus Unmasked Phase
Time Frame: 28 days for those participants wearing Dexcom G4, and 20 days for participants wearing Dexcom G6.
Measure: Mean (Standard Deviation); unit: Integer (of variation)
Arm/Group | Masked CGM Wear (Phase 1) | Unmasked CGM Wear (Phase 2)
Number analyzed (Participants) | 22 | 22
Integer (of variation) | 23.6 (5.1) | 23.0 (5.0)
Statistical Analysis 1: Comparison: Masked CGM Wear (Phase 1) vs Unmasked CGM Wear (Phase 2); Test type: Other; p = 0.25, Wilcoxon (Mann-Whitney)

14. Secondary Outcome: Mean Amplitude of Glycemic Excursion (MAGE) of Sensor Glucose Levels During Periods of CGM Wear, Masked Versus Unmasked Phase
Time Frame: 28 days for those participants wearing Dexcom G4, and 20 days for participants wearing Dexcom G6.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Masked CGM Wear (Phase 1) | Unmasked CGM Wear (Phase 2)
Number analyzed (Participants) | 22 | 22
mg/dL | 79.6 (17.8) | 74.0 (17.7)
Statistical Analysis 1: Comparison: Masked CGM Wear (Phase 1) vs Unmasked CGM Wear (Phase 2); Test type: Other; p = 0.04, Wilcoxon (Mann-Whitney)

15. Secondary Outcome: 24 Hour Continuous Overall Net Glycemic Action (CONGA) for Sensor Glucose Data During Periods of CGM Wear, Masked Versus Unmasked Phase
Description: CONGA assesses glucose variability within a predetermined time window - 24 hours in this case. Calculation of this parameter is based on the assessment of the differences between glucose values measured at regular time intervals, then on the standard deviation (SD) of these differences
Time Frame: 28 days for those participants wearing Dexcom G4, and 20 days for participants wearing Dexcom G6.
Measure: Median (Standard Deviation); unit: mg/dL
Arm/Group | Masked CGM Wear (Phase 1) | Unmasked CGM Wear (Phase 2)
Number analyzed (Participants) | 22 | 22
mg/dL | 35.6 (11.5) | 33.0 (7.0)
Statistical Analysis 1: Comparison: Masked CGM Wear (Phase 1) vs Unmasked CGM Wear (Phase 2); Test type: Other; p = 0.15, Wilcoxon (Mann-Whitney)

16. Secondary Outcome: 1 Hour Continuous Overall Net Glycemic Action (CONGA) for Sensor Glucose Data During Periods of CGM Wear, Masked Versus Unmasked Phase
Time Frame: 28 days for those participants wearing Dexcom G4, and 20 days for participants wearing Dexcom G6.
Measure: Median (Standard Deviation); unit: mg/dL
Arm/Group | Masked CGM Wear (Phase 1) | Unmasked CGM Wear (Phase 2)
Number analyzed (Participants) | 22 | 22
mg/dL | 35.5 (9.4) | 33.2 (7.1)
Statistical Analysis 1: Comparison: Masked CGM Wear (Phase 1) vs Unmasked CGM Wear (Phase 2); Test type: Other; p = 0.03, Wilcoxon (Mann-Whitney)

17. Secondary Outcome: 2 Hours, Continuous Overall Net Glycemic Action (CONGA) for Sensor Glucose Data During Periods of CGM Wear, Masked Versus Unmasked Phase
Time Frame: 28 days for those participants wearing Dexcom G4, and 20 days for participants wearing Dexcom G6.
Measure: Median (Standard Deviation); unit: mg/dL
Arm/Group | Masked CGM Wear (Phase 1) | Unmasked CGM Wear (Phase 2)
Number analyzed (Participants) | 22 | 22
mg/dL | 36.1 (11.1) | 36.9 (7.6)
Statistical Analysis 1: Comparison: Masked CGM Wear (Phase 1) vs Unmasked CGM Wear (Phase 2); Test type: Other; p = 0.04, Wilcoxon (Mann-Whitney)

18. Secondary Outcome: 4 Hours, Continuous Overall Net Glycemic Action (CONGA) for Sensor Glucose Data During Periods of CGM Wear, Masked Versus Unmasked Phase
Time Frame: 28 days for those participants wearing Dexcom G4, and 20 days for participants wearing Dexcom G6.
Measure: Median (Standard Deviation); unit: mg/dL
Arm/Group | Masked CGM Wear (Phase 1) | Unmasked CGM Wear (Phase 2)
Number analyzed (Participants) | 22 | 22
mg/dL | 38.9 (10.3) | 37.0 (6.8)
Statistical Analysis 1: Comparison: Masked CGM Wear (Phase 1) vs Unmasked CGM Wear (Phase 2); Test type: Other; p = 0.32, Wilcoxon (Mann-Whitney)

19. Secondary Outcome: Total Number of Hypoglycemic Events During the Masked Versus the Unmasked Phases of CGM Wear, as Defined by a Sensor Glucose <70 mg/dL, for at Least 15 Minutes
Description: Hypoglycemic events are defined as having glucose <70 mg/dL for at least 15 minutes, ending when glucose > the threshold. Hypoglycemic event values were normalized by dividing the number of events by the number of days of data.
Time Frame: 28 days for those participants wearing Dexcom G4, and 20 days for participants wearing Dexcom G6.
Measure: Median (Standard Deviation); unit: Number of events per period of wear
Arm/Group | Masked CGM Wear (Phase 1) | Unmasked CGM Wear (Phase 2)
Number analyzed (Participants) | 22 | 22
Number of events per period of wear | 1.6 (1.5) | 1.8 (1.3)
Statistical Analysis 1: Comparison: Masked CGM Wear (Phase 1) vs Unmasked CGM Wear (Phase 2); Test type: Other; p = 0.41, Wilcoxon (Mann-Whitney)

20. Secondary Outcome: Total Number of Hypoglycemic Events Defined by a Sensor Glucose <60 mg/dL, for at Lease 15 Minutes, During the Masked Versus Unmasked CGM Phase
Description: Hypoglycemic events are defined as having glucose <60 mg/dL for at least 15 minutes, ending when glucose > the threshold. Hypoglycemic event values were normalized by dividing the number of events by the number of days of data.
Time Frame: 28 days for those participants wearing Dexcom G4, and 20 days for participants wearing Dexcom G6.
Measure: Median (Standard Deviation); unit: Number of events per period of wear
Arm/Group | Masked CGM Wear (Phase 1) | Unmasked CGM Wear (Phase 2)
Number analyzed (Participants) | 22 | 22
Number of events per period of wear | 0.7 (0.6) | 0.5 (0.6)
Statistical Analysis 1: Comparison: Masked CGM Wear (Phase 1) vs Unmasked CGM Wear (Phase 2); Test type: Other; p = 0.04, Wilcoxon (Mann-Whitney)

21. Secondary Outcome: Total Number of Hypoglycemic Events Defined by a Sensor Glucose <54 mg/dL, for at Least 15 Minutes, During the Masked Versus Unmasked CGM Phase
Description: Hypoglycemic events are defined as having glucose <54 mg/dL for at least 15 minutes, ending when glucose > the threshold. Hypoglycemic event values were normalized by dividing the number of events by the number of days of data.
Time Frame: 28 days for those participants wearing Dexcom G4, and 20 days for participants wearing Dexcom G6.
Measure: Median (Standard Deviation); unit: Number of events per period of wear
Arm/Group | Masked CGM Wear (Phase 1) | Unmasked CGM Wear (Phase 2)
Number analyzed (Participants) | 22 | 22
Number of events per period of wear | 0.3 (0.4) | 0.2 (0.3)
Statistical Analysis 1: Comparison: Masked CGM Wear (Phase 1) vs Unmasked CGM Wear (Phase 2); Test type: Other; p = 0.08, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: For participants using a Dexcom G4 sensor, adverse event data were collected over a period of 28 days. For participants using a Dexcom G4 sensor, adverse event data were collected over a period of 20 days.
Description: Study clinicians assessed participants for adverse events at all study visits.
Arm/Group | Masked CGM Wear (Phase 1) | Unmasked CGM Wear (Phase 2)
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/23
Serious Adverse Events (participants affected / at risk) | 1/25 | 0/23
Other Adverse Events (participants affected / at risk) | 2/25 | 1/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Masked CGM Wear (Phase 1) (N=25) | Unmasked CGM Wear (Phase 2) (N=23)
Depressive episode (General disorders) | 1 (1) | 0 (0) — Episode of severe depression requiring inpatient psychiatric hospitalization.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Masked CGM Wear (Phase 1) (N=25) | Unmasked CGM Wear (Phase 2) (N=23)
Hypoglycemia requiring emergency department evaluation (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — Evaluated in the emergency department (transported from home) due to low glucose (50 mg/dL).
Skin irritation under Dexcom G4 sensor site (Skin and subcutaneous tissue disorders) | 2/13 (2) | 0/13 (0) — # At risk consists of the 13 total participants using a Dexcom G4 sensor
Mild erythema under dexcom G4 sensor adhesive (Skin and subcutaneous tissue disorders) | 1/13 (1) | 0/13 (0) — # At risk consists of the 13 total participants using a Dexcom G4 sensor
Discomfort at site of Dexcom G4 sensor (Skin and subcutaneous tissue disorders) | 1/13 (1) | 0/13 (0) — # At risk consists of the 13 total participants using a Dexcom G4 sensor

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-15): https://cdn.clinicaltrials.gov/large-docs/15/NCT03353415/Prot_SAP_000.pdf
  • Informed Consent Form (2020-07-15): https://cdn.clinicaltrials.gov/large-docs/15/NCT03353415/ICF_001.pdf